CLINICAL TRIAL: NCT02738970
Title: A Phase I, Open-Label, Two-Part, Multicenter Perjeta® Subcutaneous Dose-Finding Study in Combination With Herceptin® in Healthy Male Volunteers and Female Patients With Early Breast Cancer
Brief Title: A Dose-Finding Study of Pertuzumab (Perjeta) in Combination With Trastuzumab (Herceptin) in Healthy Male Participants and Women With Early Breast Cancer (EBC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO30185
Record Dates: First submitted 2016-03-29; First posted 2016-04-14 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Early Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Part 1-Cohort 1: Pertuzumab 420 Milligrams (mg) IV (Active Comparator): Part 1 includes healthy male participants. Participants will receive a single injection of pertuzumab 420 mg IV.
  Interventions: Drug: Pertuzumab
- Part 1-Cohort 2: Pertuzumab 400 mg SC (Experimental): Part 1 includes healthy male participants. Participants will receive a single injection of pertuzumab 400 mg SC.
  Interventions: Drug: Pertuzumab
- Part 1-Cohort 3: Pertuzumab 600 mg SC (Experimental): Part 1 includes healthy male participants. Participants will receive a single injection of pertuzumab 600 mg SC.
  Interventions: Drug: Pertuzumab
- Part 1-Cohort 4: Pertuzumab 1200 mg SC (Experimental): Part 1 includes healthy male participants. Participants will receive a single injection of pertuzumab 1200 mg SC.
  Interventions: Drug: Pertuzumab
- Part 1-Cohort 5: Trastuzumab 600 mg SC (Active Comparator): Part 1 includes healthy male participants. Participants will receive a single injection of trastuzumab 600 mg SC.
  Interventions: Drug: Trastuzumab
- Part 1-Cohort 6: Pertuzumab 400 mg SC + Trastuzumab 600 mg SC (Experimental): Part 1 includes healthy male participants. Participants will receive a single injection of co-mixed pertuzumab 400 mg and trastuzumab 600 mg SC.
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab
- Part 1-Cohort 7: Pertuzumab 1200 mg SC + Trastuzumab 600 mg SC (Experimental): Part 1 includes healthy male participants. Participants will receive a single injection of co-mixed pertuzumab 1200 mg and trastuzumab 600 mg SC.
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab
- Part 1-Cohort 8: Pertuzumab 1200 mg SC + Trastuzumab 600 mg SC (Experimental): Part 1 includes healthy male participants. Participants will receive a single injection of co-mixed pertuzumab 1200 mg and trastuzumab 600 mg SC without recombinant human hyaluronidase (rHuPH20) excipient.
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab
- Part 2-Cohort A: Pertuzumab SC + Trastuzumab SC (Experimental): Part 2 includes women with early breast cancer. Cohort A will be enrolled only if FDC of pertuzumab and trastuzumab is not feasible. Participants will receive pertuzumab and trastuzumab (600 mg) SC administered separately. The dose of pertuzumab will be identified during Part 1.
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab
- Part 2-Cohort B: Pertuzumab SC + Trastuzumab SC (Experimental): Part 2 includes women with early breast cancer. Cohorts B and C will be enrolled if FDC of pertuzumab and trastuzumab is feasible. Participants will receive pertuzumab and trastuzumab (600 mg) SC; both agents administered in one injection (co-mixed). The dose of pertuzumab will be identified during Part 1.
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab
- Part 2-Cohort C: Pertuzumab SC + Trastuzumab SC (Experimental): Part 2 includes women with early breast cancer. Cohorts B and C will be enrolled if FDC of pertuzumab and trastuzumab is feasible. Participants will receive pertuzumab and trastuzumab (600 mg) SC; both agents formulated together and administered in one injection (FDC). The dose of pertuzumab will be identified during Part 1.
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab

INTERVENTIONS:
Drug: Trastuzumab — Participants will receive a single dose of trastuzumab 600 mg SC separately, co-mixed or co-formulated with pertuzumab.
  Other Names: Herceptin, RO0452317
  Arms: Part 1-Cohort 5: Trastuzumab 600 mg SC; Part 1-Cohort 6: Pertuzumab 400 mg SC + Trastuzumab 600 mg SC; Part 1-Cohort 7: Pertuzumab 1200 mg SC + Trastuzumab 600 mg SC; Part 1-Cohort 8: Pertuzumab 1200 mg SC + Trastuzumab 600 mg SC; Part 2-Cohort A: Pertuzumab SC + Trastuzumab SC; Part 2-Cohort B: Pertuzumab SC + Trastuzumab SC; Part 2-Cohort C: Pertuzumab SC + Trastuzumab SC
Drug: Pertuzumab — Participants will receive pertuzumab as a single agent injection, co-mixed or formulated as FDC with trastuzumab depending upon cohort. The dose will range from 400 to 1200 mg.
  Other Names: Perjeta, RO4368451
  Arms: Part 1-Cohort 1: Pertuzumab 420 Milligrams (mg) IV; Part 1-Cohort 2: Pertuzumab 400 mg SC; Part 1-Cohort 3: Pertuzumab 600 mg SC; Part 1-Cohort 4: Pertuzumab 1200 mg SC; Part 1-Cohort 6: Pertuzumab 400 mg SC + Trastuzumab 600 mg SC; Part 1-Cohort 7: Pertuzumab 1200 mg SC + Trastuzumab 600 mg SC; Part 1-Cohort 8: Pertuzumab 1200 mg SC + Trastuzumab 600 mg SC; Part 2-Cohort A: Pertuzumab SC + Trastuzumab SC; Part 2-Cohort B: Pertuzumab SC + Trastuzumab SC; Part 2-Cohort C: Pertuzumab SC + Trastuzumab SC

SUMMARY:
This study involves a two-part design. Part 1 is designed to determine the optimal dose of subcutaneous (SC) Perjeta, injected alone or mixed with Herceptin, that results in comparable exposure to intravenous (IV) Perjeta. Exposure between SC Perjeta and IV Perjeta will be compared using a compilation of pharmacokinetic (PK) parameters such as area under the concentration-time curve (AUC), maximum serum concentration (Cmax), time of maximum concentration (Tmax), and serum trough concentration (Ctrough). Part 2 is designed to confirm the dosing regimen in women with EBC on the basis of safety, tolerability, and PK assessments.

ELIGIBILITY:
Inclusion Criteria:

* Part 1: Healthy male volunteers 18 to 45 years of age
* Part 1: Left ventricular ejection fraction (LVEF) at least 55 percent (%)
* Part 1: Body mass index (BMI) 18 to 32 kilograms per meter-squared (kg/m^2)
* Part 1: Normal, intact skin without tattoos or lesions in the injection area
* Part 2: Females at least 18 years of age
* Part 2: Eastern Cooperative Oncology Group (ECOG) performance status of 0
* Part 2: Previously treated, non-metastatic carcinoma of the breast
* Part 2: Baseline LVEF at least 55%
* Part 2: Negative pregnancy test and use of adequate contraceptive measures among women of childbearing potential

Exclusion Criteria:

* Part 1: Positive urine test for drugs of abuse
* Part 1: History of exposure or active viral infection of Hepatitis B, hepatitis C, or human immunodeficiency virus (HIV)
* Part 1: Cardiac disease including hypertension or hypotension
* Part 1: Lower extremity edema
* Part 1: Any clinically relevant history of systemic disease
* Part 1: History of breast cancer
* Part 1: Chronic corticosteroid use
* Part 1: Receipt of IV antibiotics within 7 days prior to enrollment
* Part 2: Concurrent malignancy requiring therapy that may interfere with pharmacokinetic investigations, or history of other malignancy within 5 years prior to Screening
* Part 2: Significant cumulative exposure to anthracyclines
* Part 2: Serious cardiac disease including uncontrolled hypertension
* Part 2: Poor hematologic, renal, or hepatic function
* Part 2: Pregnant or lactating women
* Part 2: History of exposure or active viral infection of Hepatitis B, hepatitis C, or HIV
* Part 2: Chronic corticosteroid use
* Part 2: Receipt of IV antibiotics within 7 days prior to enrollment

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2016-06-23 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration from Time Zero to Time Infinity (AUC0-inf) of Pertuzumab SC | Pre-dose (0 hours) and 6, 8, and 12 hours post-dose on Day 1; on Days 2, 3, 5, 8, 10, 15, 22, 43, 85; and at follow-up visit (up to approximately 24 months)
Maximum Serum Concentration (Cmax) of Pertuzumab SC | Pre-dose (0 hours) and 6, 8, and 12 hours post-dose on Day 1; on Days 2, 3, 5, 8, 10, 15, 22, 43, 85; and at follow-up visit (up to approximately 24 months)
Time to Reach Cmax (Tmax) of Pertuzumab SC | Pre-dose (0 hours) and 6, 8, and 12 hours post-dose on Day 1; on Days 2, 3, 5, 8, 10, 15, 22, 43, 85; and at follow-up visit (up to approximately 24 months)
Minimum Serum Concentration (Cmin) of Pertuzumab SC | Pre-dose (0 hours) and 6, 8, and 12 hours post-dose on Day 1; on Days 2, 3, 5, 8, 10, 15, 22, 43, 85; and at follow-up visit (up to approximately 24 months)
AUC0-inf of Pertuzumab IV | Pre-dose (0 hours) and 1.5 and 3 hours post-dose on Day 1; on Days 2, 3, 5, 8, 15, 22, 35, 43, 85; and at follow-up visit (up to approximately 24 months)
Cmax of Pertuzumab IV | Pre-dose (0 hours) and 1.5 and 3 hours post-dose on Day 1; on Days 2, 3, 5, 8, 15, 22, 35, 43, 85; and at follow-up visit (up to approximately 24 months)
Tmax of Pertuzumab IV | Pre-dose (0 hours) and 1.5 and 3 hours post-dose on Day 1; on Days 2, 3, 5, 8, 15, 22, 35, 43, 85; and at follow-up visit (up to approximately 24 months)
Cmin of Pertuzumab IV | Pre-dose (0 hours) and 1.5 and 3 hours post-dose on Day 1; on Days 2, 3, 5, 8, 15, 22, 35, 43, 85; and at follow-up visit (up to approximately 24 months)

SECONDARY OUTCOMES:
Percentage of Participants with Adverse Events | Baseline up to approximately 24 months
Percentage of Participants with Anti-Therapeutic Antibodies (ATAs) to Pertuzumab | Baseline, Day 22, Day 85, and 7 months post-dose (up to approximately 24 months overall)
Percentage of Participants with ATAs to Trastuzumab | Baseline, Day 22, Day 85, and 7 months post-dose (up to approximately 24 months overall)
Percentage of Participants with ATAs to rHuPH20 | Baseline, Day 22, Day 85, and 7 months post-dose (up to approximately 24 months overall)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- New Zealand (2):
  - Auckland Clinical Studies, Auckland
  - Christchurch Clinical Studies Trust, Christchurch

REFERENCES:
- [Derived] Kirschbrown WP, Wynne C, Kagedal M, Wada R, Li H, Wang B, Nijem I, Badovinac Crnjevic T, Gasser H, Heeson S, Eng-Wong J, Garg A. Development of a Subcutaneous Fixed-Dose Combination of Pertuzumab and Trastuzumab: Results From the Phase Ib Dose-Finding Study. J Clin Pharmacol. 2019 May;59(5):702-716. doi: 10.1002/jcph.1362. Epub 2018 Dec 19. PMID 30570763